CLINICAL TRIAL: NCT05788731
Title: Become of Patients From the Permanent Access to Care (PASS) in Cayenne, French Guyana, Suffering From a Chronic Disease (High Blood Pressure - Diabetes) in the Common Law Schemes
Acronym: PASSyDroit
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: PASSyDroit
Record Dates: First submitted 2023-03-08; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Access to Health Services; Health Disparity, Minority and Vulnerable Populations; Chronic Disease; Social Security
Keywords: Health care system; Vulnerable Populations; Chronic Disease; social security; French Guiana
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is an observational research, conducted at the Cayenne hospital about the future of hypertensive and/or diabetic patients after their follow-up at the Permanent Access to care (PASS). The PASS is a medico-social structure that allows access to medical monitoring and support towards common law. The main objective of the study is to evaluate the use of the common law system by these patients. Then the goal is to study the relationship between integration into the system and socio-demographic, medical characteristics, and understanding of health monitoring. Data will be collected by guided telephone interviews and the review of medical records.

DETAILED DESCRIPTION:
The problems of social inequalities in access to care are major public health issues as recalled by the Regional Health Agency (ARS) of French Guiana in the Regional Health Project (PRS). French Guiana has high precariousness indicators with half of its population living below the poverty line. In addition, health indicators are often more degraded in precarious populations. Thus, in French Guiana, there is a higher rate of premature mortality, partly attributable to obesity, sedentary lifestyle, diabetes and hypertension than in mainland France. Despite an increased need for follow-up of chronic pathologies, the precarious population faces many difficulties in accessing care. The Permanent Access to Health Care (PASS) in Cayenne is a medico-social system, created to respond to these problems. The PASS allows access to monitoring of chronic diseases and support towards the common law healthcare system. Although the phenomenon of non-use of care studied in the precarious population of western French Guiana seems primarily attributable to the absence of social security. The main objective is to evaluate the use of the common law system in hypertensive or diabetic patients treated at the PASS in Cayenne. In addition, the investigators want to study the relationship between integration into the system and the socio-demographic, medical characteristics, understanding of health monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older
* Past follow-up by the PASS of the Cayenne hospital for at least one chronic pathology identified as follows: hypertension, diabetes.
* The discharge and reorientation to general practitioner have happened between 1 month and 1 year prior to this study.

Exclusion Criteria:

* Patient with a psychiatric condition
* Refusing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Majeur patients of the PASS of CH de Cayenne with a chronic disease
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
The proportion of patients integrating the common law system | during inclusion
  It is collected through telephone interviews while inclusions are carried out.

SECONDARY OUTCOMES:
Study the relationship between system integration and socio-demographic, understanding characteristics | during inclusion
Study the relationship between system integration and medical, health follow-up | during inclusion
Proportion of patients resorting to one or more consultations with a general practitioner. | during inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Cayenne, Cayenne, French Guiana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rochemont DR, Lemenager P, Franck Y, Farhasmane A, Sabbah N, Nacher M. The epidemiology of acute coronary syndromes in French Guiana. Ann Cardiol Angeiol (Paris). 2021 Feb;70(1):7-12. doi: 10.1016/j.ancard.2020.09.032. Epub 2020 Oct 14. PMID 33067006
- See also: Samuel A, Vianney C. Les maladies chroniques touchent plus souvent les personnes modestes et réduisent davantage leur espérance de vie | Direction de la recherche, des études, de l'évaluation et des statistiques — http://drees.solidarites-sante.gouv.fr/publications-communique-de-presse/etudes-et-resultats/les-maladies-chroniques-touchent-plus-souvent
- See also: Nacher M. santé globale et guyane: étude descriptive et comparative de quelques grands indicateurs / global health and french guiana: a descriptive and comparative study of some major indicators. 24 juin 2019;10. — http://beh.santepubliquefrance.fr/beh/2020/2-3/2020_2-3_1.html
- See also: Legendre B. Le renoncement aux soins : un phénomène aux ressorts économiques mais aussi sociaux. Rev Fr Aff Soc. 2021;(3):179-204. — http://drees.solidarites-sante.gouv.fr/sites/default/files/2021-07/ER1200.pdf
- See also: Kieffer M. PrecASOG : Accès aux soins dans l'Ouest Guyanais : étude des causes de rupture thérapeutique chez les patients précaires atteints de maladie chronique. Université des Antilles; 2022 — http://theses.hal.science/tel-00134997/document